CLINICAL TRIAL: NCT05688735
Title: Prospective Randomized Vehicle-Controlled, Double-Blind Assessment of the Effect of Coconut and Sunflower Seed Oil Derived Isosorbide Diseters and Colloidial Oatmeal
Brief Title: Assessment of the Effect of Coconut and Sunflower Seed Oil Derived Isosorbide Diseters and Colloidial Oatmeal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Sytheon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDEAS_PEDS_AD
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Topical Product (Active Comparator): Topical moisturizer With Colloidal Oatmeal and Isosorbide Diesters + Topical Steroids
  Interventions: Other: Isosorbide Diester Moisturizer
- Control Topical Product (Placebo Comparator): Topical moisturizer With Colloidal Oatmeal WITHOUT Isosorbide Diesters + Topical Steroids
  Interventions: Other: Control Moisturizer

INTERVENTIONS:
Other: Isosorbide Diester Moisturizer — Isosorbide Diesters (with 0.1% colloidal oatmeal) + Topical Hydrocortisone 2.5% ointment
  Arms: Experimental Topical Product
Other: Control Moisturizer — Topical vehicle (with 0.1% colloidal oatmeal) + Topical Hydrocortisone 2.5 % ointment
  Arms: Control Topical Product

SUMMARY:
The goal of this study is to compare coconut oil and sunflower seed oil derived isosorbide disesters and colloidal oatmeal, and observe their effect on pediatric atopic dermatitis among males and females aged 2-17.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 2-17 years old at the time of consent.
* Clinical diagnosis of active atopic dermatitis
* vIGA-AD (validated Investigator Global Assessment-Atopic Dermatitis) score of "mild" (2) or "moderate" (3) at Baseline
* EASI (Eczema Area and Severity Index) score of >/= 5 at Baseline

Exclusion Criteria:

* Individuals who have a known allergy to isosorbide diesters, coconut oil, or sunflower seed oil
* Individuals who have solely hand and/or foot eczema without evidence of eczema anywhere else on their body.
* Individuals who have been on topical calcineurin inhibitors or crisaborole to the predetermined areas within two weeks of initiation of participation or unwilling to undergo a washout period.
* Subjects with an ongoing secondary infection of the skin.
* Subjects who are on systemic therapy or who need systemic therapy at the discretion of the investigator. Systemic therapies include cyclosporine, systemic steroids, methotrexate, and dupilumab. Subjects who have been on cyclosporine, systemic steroids, or methotrexate in the month prior to initiation of study intervention or are unwilling to undergo a washout period. Subjects who have been on dupilumab in two months prior to initiation of study intervention or are unwilling to undergo a washout period.
* Subjects with a diagnosis of Scabies.
* Pregnant women
* Prisoners

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | 8 Weeks
  Percent Achieving EASI 75
Itch | 8 Weeks
  Change in the Itch Visual Analog Scale from Baseline

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | 1 Week
  Change in the EASI score
Eczema Area and Severity Index (EASI) | 4 Weeks
  Change in the EASI score
Eczema Area and Severity Index (EASI) | 8 Weeks
  Change in the EASI score
Itch | 1 Week
  Change in the Itch Visual Analog Scale
Itch | 4 Weeks
  Change in the Itch Visual Analog Scale
Topical steroid use | 1 Week
  Cumulative use of topical steroid use
Topical steroid use | 4 Weeks
  Cumulative use of topical steroid use
Topical steroid use | 8 Weeks
  Cumulative use of topical steroid use
Skin Transepidermal Water Loss (TEWL) | 1 Week
  TEWL measured with a Vapometer
Skin Transepidermal Water Loss (TEWL) | 4 Weeks
  TEWL measured with a Vapometer
Skin Transepidermal Water Loss (TEWL) | 8 Weeks
  TEWL measured with a Vapometer
Skin Hydration | 1 week
  Level of skin hydration measured SkinMoistureMeterSC
Skin Hydration | 4 weeks
  Level of skin hydration measured SkinMoistureMeterSC
Skin Hydration | 8 weeks
  Level of skin hydration measured SkinMoistureMeterSC
Shift in the Skin Microbiome | 8 weeks
  Change in the relative abundance of Staphylococcus aureus on the skin

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States